CLINICAL TRIAL: NCT05184946
Title: Clinical Study of Camrelizumab Combined With SOX in the Adjuvant Treatment of Advanced Gastric Adenocarcinoma or Gastric Esophageal Junction Adenocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Shandong First Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT-002
Record Dates: First submitted 2021-12-22; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Gastric Cancer
Keywords: advanced gastric cancer, camrelizumab, adjuvant treatment
MeSH Terms: conditions — Stomach Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-PD1 combined with SOX (Experimental): Camrelizumab will be administered one day before SOX regimen.
  Interventions: Drug: Camrelizumab Combined with SOX

INTERVENTIONS:
Drug: Camrelizumab Combined with SOX — Administer camrelizumab and SOX regimen in the adjuvant treatment of advanced gastric adenocarcinoma or gastric esophageal junction adenocarcinoma
  Other Names: Anti-PD1 Combine with chemotherapy

SUMMARY:
To study the efficacy and safety of camrelizumab combined with SOX regimen for adjuvant therapy of stage III gastric cancer

DETAILED DESCRIPTION:
The purpose of this study is to explore the efficacy of anti-PD1 therapy combined with SOX for adjuvant therapy of advanced gastric cancer compared to the standard SOX regimen. Besides the efficacy, we focus on the safety and quality of life in the new treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75y, male or female; 2. Patients with gastric adenocarcinoma or gastroesophageal junction adenocarcinoma confirmed by histology or cytology; 3. Patients with stage III gastric adenocarcinoma or gastroesophageal junction adenocarcinoma who have not received any antitumor therapy besides surgery; 4. ECOG score: 0 ~ 1; 5. Expected survival ≥12 weeks; 6. The main organs function are well, and the laboratory test data meets the following standards: (1) Blood routine: neutrophil absolute count ≥1.5×109/L (or greater than the lower limit of laboratory normal value in the research center), platelet count ≥100×109/L, hemoglobin ≥90g/L; (2) Liver function: serum total bilirubin ≤1.5 times the upper limit of standard value (ULN), AST and ALT≤2.5 times ULN, and ≤5 times ULN if liver metastasis exists; (3) Renal function: CrCl≥ 60mL /min/1.73m2 (calculated according to the Cockcroft-Gault formula); 7. Female subjects with the fertility, as well as the partner of male subjects with the fertility, need to use an approved medical contraception (such as intrauterine device, the pill or condoms) during the research and at least 6 months from the last treatment of camrelizumab or chemotherapy; 8. HER2 negative, volunteering to provide tumor tissue samples after surgery and adjuvant therapy; 9. Voluntarily participated in the study and signed informed consent with good compliance and follow-up.

Exclusion Criteria:

1. History of gastrointestinal perforation and/or fistula within 6 months prior to first medication; 2. Uncontrolled pleural effusion, pericardial effusion or peritoneal effusion requiring repeated drainage; 3. Allergic to carrelizumab, oxaliplatin, or tegio; 4. Received any of the following treatments: a. Enrolled in another clinical study at the same time; b. Prior to initial use of the study drug, antitumor therapy (including radiotherapy, chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biotherapy, or tumor embolization, etc.) was performed; c. Subjects requiring corticosteroids (> 10mg prednisone equivalent daily dose) within 2 weeks prior to initial use of the study drug. Other special situations require communication with the researcher. In the absence of active autoimmune disease, inhaled or topical steroids and adrenocorticosteroid replacement at doses > 10mg/d of prednisone efficacy are permitted; d. Those who have received antitumor vaccine or have received live vaccine within 4 weeks prior to the first administration of the study drug; e. Major surgery or severe trauma within 4 weeks prior to first use of the study drug; 5. Patients with central nervous system metastasis; 6. Have active autoimmune diseases or a history of autoimmune diseases (such as interstitial pneumonia, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to the above diseases or syndromes); Except for patients with epilepsy or recovered childhood asthma/allergy without any intervention as adults; Autoimmune mediated hypothyroidism treated with stable doses of thyroid replacement hormone; Type 1 diabetes with a steady dose of insulin; 7. Have a history of immunodeficiency, including HIV positive, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation and allogeneic bone marrow transplantation, or active hepatitis (hepatitis b: HBV-dna test value over 500IU/ml or 2500 copies /ml); 8. The subject has cardiovascular clinical symptoms or diseases that are not well controlled, including but not limited to: e.g. : (1) NYHA class II or higher heart failure; (2) unstable angina; (3) myocardial infarction occurred within 1 year; (4) Clinically significant supraventricular or ventricular arrhythmias are still poorly controlled without or after clinical intervention; 9. Severe infection (CTCAE5.0 > 2) occurred within 4 weeks prior to the first use of the study drug, such as severe pneumonia, bacteremia, and infection complications requiring hospitalization; Baseline chest imaging suggests active lung inflammation, signs and symptoms of infection within 2 weeks prior to initial use of the study drug, or the need for oral or intravenous antibiotic treatment, except for prophylactic use of antibiotics; 10. A history of interstitial lung disease (excluding radiation pneumonia or non-infectious pneumonia without hormone therapy); 11. Patients with active tuberculosis infection found by history or CT examination, or patients with active tuberculosis infection history within 1 year before enrollment, or patients with active tuberculosis infection history more than 1 year ago but without formal treatment;12. Diagnosis of any other malignancy, other than malignancies with a low risk of metastasis and death (5-year survival > 90%), such as adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix, within 5 years prior to first use of the study drug; 13. Pregnant or lactating women; 14. In the judgment of the investigator, the subject has other factors that may cause him/her to be forced to terminate the study, such as other serious diseases (including mental illness) requiring combined treatment, seriously abnormal laboratory test values, family or social factors that may affect the safety of the subject or the collection of test data; 15. According to the investigator's judgment, subjects have other factors that may cause them to be forced to terminate the study, such as other serious diseases (including mental illness) requiring combined treatment, seriously abnormal laboratory test values, family or social factors that may affect subjects' safety or the collection of test data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-10-09 (Actual); Primary Completion 2025-10-08 (Estimated); Study Completion 2025-10-08 (Estimated)

PRIMARY OUTCOMES:
3 years disease free survival rate | 3 years
  With 3 years of follow-up,the three-year disease-free survival rate will be observed and compared with the target value.

SECONDARY OUTCOMES:
overall survival time | 2 years, 3 years
  With 2 and 3 years of follow-up,the 2/3-year overall survival time will be observed and compared with the target value.

CONTACTS AND LOCATIONS:
Overall Officials: Haiyan liu, Principal Investigator — The Second Affiliated Hospital of Shandong First Medical University
Locations (1):
- The Second Affiliated Hospital of Shandong First Medical University, Tai’an, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Janjigian YY, Shitara K, Moehler M, Garrido M, Salman P, Shen L, Wyrwicz L, Yamaguchi K, Skoczylas T, Campos Bragagnoli A, Liu T, Schenker M, Yanez P, Tehfe M, Kowalyszyn R, Karamouzis MV, Bruges R, Zander T, Pazo-Cid R, Hitre E, Feeney K, Cleary JM, Poulart V, Cullen D, Lei M, Xiao H, Kondo K, Li M, Ajani JA. First-line nivolumab plus chemotherapy versus chemotherapy alone for advanced gastric, gastro-oesophageal junction, and oesophageal adenocarcinoma (CheckMate 649): a randomised, open-label, phase 3 trial. Lancet. 2021 Jul 3;398(10294):27-40. doi: 10.1016/S0140-6736(21)00797-2. Epub 2021 Jun 5. PMID 34102137
- [Background] Hermann RM, Christiansen H. [A new standard is emerging: PD-1 maintenance therapy after neoadjuvant radiochemotherapy and curative resection of oesophageal and AEG carcinomas (CheckMate 577)]. Strahlenther Onkol. 2021 Nov;197(11):1040-1042. doi: 10.1007/s00066-021-01849-3. Epub 2021 Sep 13. No abstract available. German. PMID 34515819